CLINICAL TRIAL: NCT00351156
Title: A Multicenter Study to Evaluate and Characterize the Ex Vivo Effect of Pharmacological Chaperone Therapy in Blood Cell Lines Derived From Patients With Gaucher Disease
Brief Title: Study to Evaluate Blood Cell Lines From Patients With Gaucher Disease
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Other Study IDs: GAU-CL-001
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Gaucher Disease
Keywords: Gaucher Disease; Gaucher Disease, Type 1; Gaucher Disease, Type 2; Gaucher Disease, Type 3; Neuronopathic Gaucher Disease; Non-Neuronopathic Gaucher Disease; Lysosomal Storage Disease; Metabolism, Inborn Errors; Metabolic Diseases; Sphingolipidoses; Genetic Diseases, Inborn
MeSH Terms: conditions — Gaucher Disease; Lysosomal Storage Diseases; Metabolism, Inborn Errors; Metabolic Diseases; Sphingolipidoses; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood

INTERVENTIONS:
Procedure: Blood sample

SUMMARY:
The purpose of this study is to learn more about Gaucher disease. The information we collect from medical histories and a blood sample from people with Gaucher disease may help us pinpoint certain things that are different between people who have Gaucher disease and people who do not have Gaucher disease. This information may be useful in the future to help find new treatments for Gaucher disease.

DETAILED DESCRIPTION:
This study is designed to evaluate the ex vivo response to pharmacological chaperone therapy by testing blood samples from previously treated and untreated patients with Gaucher disease. The study will include patients with non-neuropathic Gaucher disease (type I) and neuropathic Gaucher disease (types II and/or III).

All subjects will participate in one study visit. Clinical information will be collected retrospectively from medical records. Information collected will include Gaucher disease diagnosis and history, medical history, family history, assessments of clinical severity, and genotype. A blood sample will be collected and various cells will be isolated for laboratory testing and research.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent by subject or legal guardian
2. Male or female of any age
3. Confirmed diagnosis of Gaucher disease with known genotype
4. Clinically stable and either treatment naïve or on a stable dose of enzyme replacement therapy and/or substrate reduction therapy for at least 6 months prior to study entry
5. Available medical records for collection of retrospective clinical information

Exclusion Criteria:

1. Received any investigational product within 30 days prior to study entry
2. Other significant disease or be otherwise unsuitable for the study, as determined by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Gaucher disease
Sampling Method: Non-Probability Sample
Enrollment: 50
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ludwig, M.D., Study Director — Amicus Therapeutics, Inc.
Locations (7):
- United States (7):
  - University of California - San Francisco, San Francisco, California
  - University Research Foundation for Lysosomal Storage Diseases, Inc., Coral Springs, Florida
  - Emory University Lysosomal Storage Disease Center, Decatur, Georgia
  - National Institute of Neurological Disorders and Stroke, NIH, Bethesda, Maryland
  - New York University School of Medicine, Neurogenetics Department, New York, New York
  - Lysosomal Disease Center, Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania